CLINICAL TRIAL: NCT04323267
Title: Efficacy of Digital Home-Exercise Therapy Application For Patients With Non-Surgical Knee Injuries: A Randomized, Controlled Trial
Brief Title: Digital Home-Exercise Therapy Application For Patients With Non-Surgical Knee Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jacob L. Sellon, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-007031
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Knee Injuries; Knee Osteoarthritis; Patellofemoral Syndrome
Keywords: knee pain; knee osteoarthritis; patellofemoral syndrome; physical therapy; digital health
MeSH Terms: conditions — Knee Injuries; Osteoarthritis, Knee; Patellofemoral Pain Syndrome | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Home Exercise Program (Experimental): Limber Digital Application Device (3 x a week for 8 weeks)
  Interventions: Device: Limber Digital Application
- Physical therapy (Active Comparator): Therapy prescription 2 x a week for 8 weeks (specified by physician)
  Interventions: Behavioral: Physical therapy Therapy

INTERVENTIONS:
Device: Limber Digital Application — A mobile application was recently developed to address these needs. The application provides evidence-based, symptom specific home-exercise video programs for MSK conditions, as well as clinically-validated outcome measures for tracking progress.
  Arms: Digital Home Exercise Program
Behavioral: Physical therapy Therapy — Therapy prescription 2 x a week for 8 weeks (specified by physician)
  Arms: Physical therapy

SUMMARY:
Knee pain is one of the most prevalent musculoskeletal disorders in the United States. Conservative treatments generally consist of pharmacological agents and physical therapy. Unfortunately, such conservative care is often mismanaged, and little data is collected on clinical outcomes. The proposed investigation utilizes a novel and state-of-the-art mobile application (DETP) to guide an at-home exercise therapy program for non-operative knee pain. The purpose of this study is conducting a single-blind randomized, controlled, superiority study to compare the DETP to conventional physical therapy (PT). The investigators will seek to determine improvement in pain and function in PROMIS measures as the primary outcome. The investigators will also evaluate satisfaction with the application as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75, inclusive.
* Diagnosis of knee injury. For participants enrolled from the Mayo healthcare system database, knee injury identified from electronic medical records.
* Pain Numerical Rating Scale score of 4 or greater on a 0-10 scale (0 = no pain, 10 = pain).
* Participants must be diagnosed with a knee injury and the next step of care is either a home exercise program or external physical therapy ordered at the academic center.
* Prescribed external physical therapy (i.e., therapy not completed at Mayo Clinic in Rochester/Minneapolis).

Exclusion Criteria:

* No access to android or iPhone smartphone
* BMI greater than or equal to 35
* Previously completed series of physical therapy visits for knee injury within the past 12 months for the same injury (received one introduction PT session as seen in executive program will not be considered an exclusion).
* Recommended by a physician for consideration of total knee replacement.
* Diagnosis of rheumatoid arthritis, fibromyalgia, gout in the knee, or other systemic rheumatic disease.
* Hospitalization for a stroke, heart attack, heart failure, or had surgery for blocked arteries in the past 12 months.
* Total joint replacement knee surgery, bucket-handle meniscus tear, ACL tear, or other knee surgery in the past 12 months.
* Unable to speak English.
* Active diagnosis of psychosis.
* Fall history deemed by a physician to impose risk for potential injury with participation in a home-based exercise program.
* Severely impaired hearing or speech.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Score | 8 weeks
  Pain is measured by 0-100. 0 = no pain and 100 = very high pain
PROMIS Physical Function CAT | 8 weeks
  Function is measured by 0-100. 0= no function and 100 = high function

SECONDARY OUTCOMES:
Subject Satisfaction Questions | 8 weeks
  Satisfaction questions

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sellon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials